CLINICAL TRIAL: NCT01314014
Title: A Phase II Study of Amplimexon® (Imexon for Injection) for the Treatment of Previously Treated Follicular and Aggressive Lymphoma in Adults
Brief Title: Imexon for Relapsed Follicular and Aggressive Lymphomas
Acronym: ULYM11011
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: University of Arizona (Other)
Responsible Party: Principal Investigator, Paul Barr, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 36191
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2015-12

CONDITIONS: Follicular Lymphoma; Small Lymphocytic Lymphoma; Marginal Zone Lymphoma; Lymphoplasmacytic Lymphoma; Diffuse Large B Cell Lymphoma; Mantle Cell Lymphoma; Burkitt's Lymphoma
Keywords: Non Hodgkin's Lymphoma; Lymphoma, Low Grade; Lymphoma, Intermediate Grade; Lymphoma, High Grade; Lymphoma, B Cell
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Burkitt Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — 4-imino-1,3-diazabicyclo(3.1.0)hexan-2-one; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imexon (Experimental): Subjects will be treated on Days 1-5 of 21-day treatment cycles for up to one year. Following pre-treatment with anti-emetics Amplimexon will be given by intravenous infusion over 60 minutes.
  Interventions: Drug: Imexon

INTERVENTIONS:
Drug: Imexon — Amplimexon will be administered daily on Days 1-5 of 21-day treatment cycles as an intravenous infusion over a time course of 60 minutes. Subjects will receive 17 cycles of therapy for a total of one year on treatment. The Amplimexon starting dose for each subject in this study is 1000 mg/m² on each treatment day. Dose may be reduced by 25% for toxicity; after 2 dose reductions, subjects must be withdrawn from treatment.
  Other Names: Amplimexon (imexon for injection)

SUMMARY:
The purpose of this study is to determine whether Amplimexon (imexon for injection) is effective in the treatment of indolent and aggressive lymphomas that have progressed after treatment with standard therapies.

DETAILED DESCRIPTION:
A phase II exploratory trial of imexon in lymphoma is justified by: (1) the observation of clinical activity (partial response to the drug observed in phase I testing in a subject with refractory indolent lymphoma); (2) the finding that imexon prevents the development of human immunoblastic lymphoma in SCID mice; (3) the finding that lymphoma cell lines are killed by readily achievable doses; and (4) translational studies implicating the importance of the redox state of the cancer cell.

The dose and schedule chosen (1000 mg/m2 daily X 5 days every 3 weeks) is based on tolerability and subject acceptance in prior AmpliMed phase I studies.

The planned correlative studies should help to identify potential biomarkers for response to imexon and provide further insight into potential mechanisms of imexon action hypothesized from results of prior laboratory studies.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis:

   Group 1: Histologically confirmed indolent NHL, including follicular (any grade), small lymphocytic lymphoma, marginal zone lymphoma and lymphoplasmacytic lymphomaGroup 2: histologically confirmed diffuse large B-cell, mantle cell, Burkitt, Burkitt-like, and diffuse large B-cell transformed from indolent non-Hodgkin's lymphoma.
2. Prior treatment:

   Group 1: (indolent histologies): Patients must have demonstrated relapsed or refractory disease to 1 prior treatment regimen. The maximum number of prior regimens used for treatment is not specified.

   Group 2: (aggressive histologies): Patients must have demonstrated relapsed or refractory disease to at least 1 prior treatment regimen. In the case of de novo diffuse large B-cell lymphoma, prior treatment must include R-CHOP or R-CHOP-like therapy, as well as second line autologous stem cell transplantation unless the patient is not eligible. The maximum number of prior regimens is not specified.
3. At least one target lesion, measurable by radiographic methods according to the 2007 Revised Response Criteria for Malignant Lymphoma.
4. ECOG Performance Status 0-2.
5. No clinical or laboratory evidence of central nervous system disease.
6. Adult (age 18 years or older).
7. Projected life expectancy >4 months.
8. If female, neither pregnant (negative pregnancy test required at screening) nor lactating.
9. If of child-bearing potential, must be able to use and agree to use medically acceptable contraception for the duration of the study. For female subjects who are neither post-menopausal nor surgically sterilized, this includes oral or injectable hormonal methods, barrier methods such as an intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence. Male subjects must also agree to use an acceptable method for contraception for the duration of the study.
10. No major infection or serious uncontrolled concomitant disease. Fully recovered from any major surgery.
11. No evidence of other concurrent active malignancy.
12. At least 4 weeks since any prior cancer chemotherapy (2 weeks for corticosteroids), antibody therapy, or radiotherapy.
13. Prior radiotherapy to less than an estimated 25% of the bone marrow. In addition, the target lesion(s) must not have been previously irradiated.
14. Clinical laboratory values within the following limits:

    1. Hgb >/=10.0 g/dL
    2. Absolute neutrophil count ANC >/=1,500/mm3
    3. Platelets >/=75,000/mm3
    4. Serum creatinine </=2.0 times upper limit of normal
    5. Serum bilirubin </=2.0 times upper limit of normal
    6. Serum AST and ALT </=3 times upper limit of normal
15. G6PD level >/= lower limit of normal
16. Able and willing to render informed consent and to follow protocol requirements.

Exclusion Criteria:

1. Diagnosis of lymphoma based on fine needle aspirate.
2. Curative therapy is indicated or possible.
3. Absence of a measurable target lesion, or the only target lesion was previously irradiated.
4. Symptoms, exam findings, or laboratory findings to suggest central nervous system disease involvement.
5. Age < 18 years
6. Projected life expectancy <4 months.
7. Pregnant or lactating.
8. Unable or unwilling to use medically acceptable contraception, if of childbearing potential.
9. Evidence of major infection or other serious uncontrolled concomitant illness. Not fully recovered from prior major surgery.
10. Evidence of other active malignancy.
11. Prior radiotherapy, antibody therapy, or cancer chemotherapy within 4 weeks before start of treatment (2 weeks for corticosteroids). Prior radiotherapy to >25% of the bone marrow.
12. Clinical laboratory values outside of permitted ranges.
13. Respiratory insufficiency requiring oxygen therapy; angina at rest, or myocardial infarction in previous 3 months; history of life threatening ventricular arrhythmia; uncompensated CHF or NYHA Grade 3 or 4 cardiac disease.
14. Unable or unwilling to give informed consent and to follow protocol requirements.
15. Failure to meet any of the eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-05; Primary Completion 2013-03 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Barr, MD, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - Arizona Cancer Center, University of Arizona, Tucson, Arizona
  - University of Rochester Medical Center, Rochester, New York

REFERENCES:
- [Result] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Derived] Barr PM, Miller TP, Friedberg JW, Peterson DR, Baran AM, Herr M, Spier CM, Cui H, Roe DJ, Persky DO, Casulo C, Littleton J, Schwartz M, Puvvada S, Landowski TH, Rimsza LM, Dorr RT, Fisher RI, Bernstein SH, Briehl MM. Phase 2 study of imexon, a prooxidant molecule, in relapsed and refractory B-cell non-Hodgkin lymphoma. Blood. 2014 Aug 21;124(8):1259-65. doi: 10.1182/blood-2014-04-570044. Epub 2014 Jul 11. PMID 25016003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study occured at two academic medical centers (University of Rochester and Arizona Cancer Center) from June 7, 2011 through March 4, 2013.
Period: Overall Study
Arm/Group | Imexon
Started | 22
Completed | 22 (Treatment continued for as long as the subject derived benefit.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Imexon
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 64 [43 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate of of Participants to Imexon in the Treatment of Relapsed/Refractory Indolent and Aggressive Lymphomas
Description: CT, PET, or MRI scans for the assessment of objective tumor responses were performed at baseline, after cycle 2, and every 3 cycles thereafter until disease progression. Standard response criteria from the International Harmonization Project on Lymphoma were used for classification of objective tumor responses. Response was defined as PR (Regression of measuable disease and no new sites) if >= 50% decrease in sum of the product of the diameters of up to 6 largest dominant masses; no increase in size of other nodes (a) [18F]fluorodeoxyglucose (FDG)-avid or PET prior to therapy; one or more (PET) positive at previously involved site (b) Variably FDG-avid or PET negative; regression on CT.
Time Frame: One year
Population: 20 subjects were evaluable for response, 2 subjects discontinued therapy during cycle 1 due to progressive disease and grade 5 sepsis respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Imexon
Number analyzed (Participants) | 20
percentage of participants | 30 [9.9 to 50.1]

2. Secondary Outcome: Median Time to Progression Free Survival in Participants With Relapsed/Refractory Indolent and Aggressive Lymphomas
Description: Measured from start of treatment until disease progression or death from any cause.
Time Frame: up to 25 months
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Imexon
Number analyzed (Participants) | 20
months | 2.4 [1.2 to 9.0]

ADVERSE EVENTS:
Time Frame: From first dose of study treatment through 30 days after last dose.
Description: For each subject, AE recording began on Day 1 of the first treatment cycle, and continued until the subject completed the protocol or withdrew from the study for any reason. AEs were followed clinically until they resolved or 30 days after the last dose of study drug was received, whichever occured first.
Arm/Group | Imexon
Serious Adverse Events (participants affected / at risk) | 9/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imexon (N=22)
Vomiting (Gastrointestinal disorders) | 2 (2)
Bronchial infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Renal and urinary disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imexon (N=22)
Fatigue (General disorders) | 20 (26)
Diarrhea (Gastrointestinal disorders) | 16 (28)
Nausea (Gastrointestinal disorders) | 15 (23)
Anemia (Blood and lymphatic system disorders) | 11 (29)
Fever (General disorders) | 10 (14)
Constipation (Gastrointestinal disorders) | 9 (11)
White blood cell decreased (Blood and lymphatic system disorders) | 8 (14)
Platelet count decreased (Blood and lymphatic system disorders) | 8 (19)
Vomiting (Gastrointestinal disorders) | 6 (7)
Anorexia (Metabolism and nutrition disorders) | 8 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Chills (General disorders) | 7 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (11)
Neutrophil count decreased (Investigations) | 5 (18)
Respiratory infection (Infections and infestations) | 4 (6)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Hypotension (Vascular disorders) | 4 (4)
Weight loss (Investigations) | 5 (7)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Headache (Nervous system disorders) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Creatinine increased (Investigations) | 3 (4)
Dysgeusia (Nervous system disorders) | 4 (4)
Malaise (General disorders) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (7)
Edema limbs (General disorders) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)
Insomnia (Psychiatric disorders) | 3 (3)
Paresthesia (Nervous system disorders) | 3 (4)
Oral dysesthesia (Gastrointestinal disorders) | 3 (3)
Alanine aminotransferase increased (Investigations) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No